CLINICAL TRIAL: NCT05415852
Title: Comparison Between Different Types of LASER in the Treatment of Onychomycosis, a Randomized Controlled Trial
Brief Title: Lasers in Onychomycosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar El Sayed, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Lasers in onychomycosis
Record Dates: First submitted 2022-05-20; First posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis | interventions — Lasers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- fractional CO2 laser (Active Comparator): Laser
  Interventions: Device: Laser
- Pulsed dye laser (Active Comparator): Laser
  Interventions: Device: Laser
- Nd Yag (Active Comparator): Laser
  Interventions: Device: Laser
- Q switched Nd Yag (Active Comparator): Laser
  Interventions: Device: Laser

INTERVENTIONS:
Device: Laser — Laser

SUMMARY:
Onychomycosis is the most common nail disease, representing more than 50% of all onychopathies. Future studies on the absorption spectra of dermatophyte fungi will be needed to develop lasers that effectively exploit absorption differences in fungi and dermal tissue.

DETAILED DESCRIPTION:
Treatments with antifungals may not be successful due to several factors, including the long time required to apply topical medications, the side effects of systemic drugs, and the application of insufficient medication to the target area. Even with adequate systemic or topical therapy, the persistence of fungal infections is not uncommon. In light of these limitations, laser therapy has been proposed as an alternative option for onychomycosis therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with onychomycosis.

Exclusion Criteria:

* Patients with excessive manual work

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-25 (Estimated); Primary Completion 2022-09-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Onychomycosis severity index | change from baseline at 3 months
  clinical assessment